CLINICAL TRIAL: NCT01872637
Title: Improving Activity, Participation And Function After Acute Hospitalization In Older Adults With Multiple Chronic Conditions: Phase II Randomized Controlled Trial
Brief Title: Improving Function, Participation and Function After Acute Hospitalization in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Arcadia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0432; Innovator's Fund (Other Grant/Funding Number: Abington Memorial Innovator's Fund); APTA (Other Grant/Funding Number: APTA Home Health Section)
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Frail Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Multi-Component Intervention (Experimental): Patients in this exercise group will receive 10-18, 45-60 minute, physical therapy visits in their home. This group will consist of progressive resistance exercises for the upper and lower extremity with a portable training device, a motor control-based program of gait/balance training, Activities of Daily Living (ADL) training, and mobility training.
  Interventions: Behavioral: Progressive Multi-Component Intervention
- Usual Care Group (Active Comparator): The patients in this group will receive approximately five visits of "usual home care" but the total number of visits will be determined by the therapist as part of usual care. These visits will likely occur at 1-2 times per week for 3-4 weeks. This group will receive intervention as determined by the physical therapist's initial examination. Interventions may include patient education, home exercises, low intensity strengthening exercise, training in gait, balance and transfers; home safety and assistive device assessment.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Progressive Multi-Component Intervention
  Arms: Progressive Multi-Component Intervention
Behavioral: Usual Care
  Arms: Usual Care Group

SUMMARY:
Hospitalization increases the risk for new disability in older adults. In the current health care system, home health physical therapy is understudied and often does not return older adults to prior levels of function. The proposed evidence-based multicomponent intervention that combines high intensity strength training and motor control based systems of gait and balance training will advance clinical practice by providing an intervention strategy for practitioners. If successful, improving patient function and decreasing re-hospitalization rates and falls will have large cost saving implications.

DETAILED DESCRIPTION:
Background: Hospitalized older adults are 59.8 times more likely to develop disability than those who are not hospitalized. No studies have examined the effectiveness of Home Health (HH) physical therapy on improving function in older adults with multiple co-morbidities after hospitalization. Our goal is to enable older adults with multiple chronic conditions to recover function by providing adequate content and dose of intervention after hospitalization. This intervention is designed to work within the existing Medicare system and has potential for immediate clinical impact.

Purpose: The primary aim of our study is to determine if a progressive multi-component (PMC) intervention, initiated upon discharge from an acute care hospital, improves gait speed at the end of one 60-day episode of care, more than documented usual care (UC) physical therapy. We hypothesize that there will be a greater improvement in gait speed measured for the PMC group compared to the UC group following one episode of care. Benefits of PMC will be apparent at the end of usual care and will increase further at the end of the 60 day episode of care (primary endpoint).

Design: We propose to conduct a single blind randomized two arm clinical trial (RCT) in older adults discharged from acute care and referred to HH physical therapy. Both interventions (PMC & UC) will be Medicare-reimbursed. All assessments and interventions will occur in the patients' homes.

Methods: Twenty individuals who are 65 years of age or older with multiple co-morbid conditions will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* referred to home care physical therapy
* have at least 3 comorbid conditions
* ambulatory without human assistance prior to hospitalization

Exclusion Criteria:

* acute lower extremity fractures with weight-bearing restriction
* elective joint replacement surgery
* active cancer diagnosis
* acute cardiac surgery
* lower extremity amputation
* referred to hospice home health physical therapy
* dialysis
* hospice care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Gait Speed | 60 days
  Time it takes to walk a 4 meter path, key to independent functioning

SECONDARY OUTCOMES:
Modified Physical Performance Test (mPPT) | 60 days
  Assesses 7 different tasks. Based on the time taken to complete the tasks, a score from 0 (unable to complete) to 4 (performed quickly and easily) if given for each task. A maximal score of 28 is given, including tasks that involved the upper and lower extremity function.
Late-Life Function and Disability Instrument (LLFDI) | 60 days
  Evaluates limitation and frequency of taking part in 16 major life tasks in its disability component, and 32 functional tasks in its functional component, of which 14 tasks comprise basic lower extremity function.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Stevens-Lapsley, PT, PhD, Principal Investigator — University of Colorado, Denver; Kate Mangione, PT, PhD, Principal Investigator — Arcadia University
Locations (2):
- United States (2):
  - University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado
  - Arcadia University, Glenside, Pennsylvania